CLINICAL TRIAL: NCT06559787
Title: Volumetric Quantification of Epicardial Fat Using Semiautomated High Resolution Atrial CT Segmentation in Patients With Atrial Fibrillation Receiving Catheter Ablation
Acronym: AFAT
Status: Active, not recruiting | Type: Observational
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: The German Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: AFAT-Studie
Record Dates: First submitted 2024-07-09; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Atrial Fibrillation
Keywords: epicardial fal
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this prospective observational study is to learn about the influence of epicardial fat on the success of catheter ablation in patients with atrial fibrillation.

DETAILED DESCRIPTION:
A volumetric quantification of epicardial fat is examined by dual source cardiac computet tomography in patients with paroxysmal or persistent atrial fibrillation prior to receiving their first catheter ablation for atrial fibrillation. After ablation the recurrence of arrhythmia is examined after 3 and 6 months respectively.

ELIGIBILITY:
Inclusion Criteria:

* patients with planned catheter ablation due to paroxysmal or persistent atrial fibrillation
* written informed consent
* planned computet tomography

Exclusion Criteria:

* history of left atrial catheter ablation
* minor patients or patients not capable of giving written informed consent
* contraindication for computet tomography with contrast agents (e.g. allergy to contrast agents or relevant renal insufficiency or hyperthyreosis)
* patients with congenital heart defects or history of cardial surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: at least 200 patients planned
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-08-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Influence of epicardial adipose tissue (EAT) volume on 1 year arrhythmia recurrences after catheter ablation | measurement of epicardial fat at baseline; anamnestic and ECG-control of arrhythmia after 3, 6 and 12 months
  influence of EAT volume quantified by volumetric CT segmentation on 1 year arrhythmia recurrences after catheter ablation for paraxysmal or persistent atrial fibrillation

SECONDARY OUTCOMES:
associations between EAT and gender, BMI, cholesterol levels, body fat | measurement of epicardial fat at baseline; anamnestic and ECG-control of arrhythmia after 3, 6 and 12 months
  associations between EAT and gender, BMI, cholesterol levels, body fat
associations between EAT and left atrial wall thining | measurement of epicardial fat at baseline; anamnestic and ECG-control of arrhythmia after 3, 6 and 12 months
  associations between EAT and left atrial wall thining
associations between EAT and low voltage areas quantified by high density electroanatomical mapping | measurement of epicardial fat and catheter ablation at baseline
  associations between EAT and low voltage areas quantified by high density electroanatomical mapping

CONTACTS AND LOCATIONS:
Overall Officials: Nico Erhard, Dr. med., Principal Investigator — Deutsches Herzzentrum München
Locations (1):
- Deutsches Herzzentrum, München, Germany

REFERENCES:
- [Derived] Englert F, Obermeyer T, Bahlke F, Popa M, Krafft H, Martinez AT, Syvari J, Tydecks M, Dischel D, Koops E, Reiter T, Telishevska M, Lengauer S, Bressem K, Hadamitzky M, Hessling G, Deisenhofer I, Erhard N. Epicardial adipose tissue and ablation outcomes in obese patients with paroxysmal atrial fibrillation: A comparison of pulsed field and radiofrequency ablation. Heart Rhythm O2. 2025 Sep 25;6(12):1901-1910. doi: 10.1016/j.hroo.2025.09.020. eCollection 2025 Dec. PMID 41541734